CLINICAL TRIAL: NCT05580874
Title: Investigation of the Effect of Massage on Stress Behaviors and Salivary Cortisol Levels in Premature Babies
Brief Title: The Effect of Massage on Stress in Premature Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Tepecik Training and Research Hospital (Other); Ege University (Other)
Responsible Party: Principal Investigator, Pınar Dogan, RN, MSc, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-1.1T/54
Record Dates: First submitted 2022-06-30; First posted 2022-10-14 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Stress; Cortisol
Keywords: Massage; Premature; Stress
MeSH Terms: conditions — Premature Birth | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage group (Experimental): Infants in the massage group received a ten-minute massage once a day, one hour after the morning feeding (between 9.30-11.30 am). Video recordings were made to observe the stress behaviors of the infants before, during and after the massage. Vital signs will be recorded a minute before the starting of the massage, at fifth minutes during the procedure and a minute after the end of the massage, and a video will be recorded during these processes. A saliva cortisol sample will be taken the massage five minutes before and 30 minutes after the massage. The scores given to the "Newborn Stress Scale" will be evaluated by watching the videos recorded after the procedure by experts in the field.
  Interventions: Other: Massage
- Control group (Other): Infants in the swaddling group will form the control group. The swaddling process will be done one hour after the babies are feding (between 9.30-11.30 am). Before, during and after the swaddling procedure, the video will be recorded to observe the stress behavior of the babies. A minute before swaddling, video recording will start. Infants will be swaddling for ten minutes and video recording will be continue. After this process, a minute video recording will be made while the baby is not swaddling. Vital signs will be recorded one minute before starting the swaddling at fifth minutes during the procedure, and a minute after the swaddling.
  A saliva cortisol sample will be taken five minutes before and 30 minutes after the swaddling. The scores given to the "Newborn Stress Scale" will be evaluated by watching the videos recorded after the procedure by experts in the field.
  Interventions: Other: Swaddling

INTERVENTIONS:
Other: Massage — The babies in the massage group were given a massage once a day.
  Arms: Massage group
Other: Swaddling — Control group
  Arms: Control group

SUMMARY:
The practices of the neonatal intensive care unit that reduce the stress of premature babies and respond to behavioral cues have a positive effect on the development of newborns. The stress experienced by premature infants affects the baby's behavior and laboratory findings. Massage is an effective application in facilitating the adaptation of premature babies to extrauterine life and ensuring that they are least affected by adverse environmental conditions. Massage in premature babies has an important place in reducing stress and supporting psychological, mental and physiological development as a healthy tactile stimulus.

DETAILED DESCRIPTION:
This study was planned to examine the effects of massage on stress behaviors and salivary cortisol levels in premature infants. The research was planned on a randomized controlled experimental. In the research, the group to which massage will be procedure is the experimental group, and the group to which the swaddling procedure will be the control group will form.

ELIGIBILITY:
Inclusion Criteria:

* Families being voluntary to participate in the study
* Babies being born between 30 and 36 weeks plus 6 days of gestation
* Postnatal 3-5. premature babies between days
* Not taking analgesics or sedatives
* Absence of congenital anomaly
* Absence of skin disease
* The premature babies passing to oral feeding
* Not having a proven sepsis diagnosis
* No need for mechanical ventilator support

Exclusion Criteria:

* Having a congenital anomaly
* Presence of skin disease
* Having intracranial bleeding
* Having sepsis
* Receiving phototherapy
* Taking analgesic / sedative type drugs

Ages: 30 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol levels | 5 minutes before massage
Salivary cortisol levels | 5 minutes before swaddling
Salivary cortisol levels | 30 minutes after massage
Salivary cortisol levels | 30 minutes after swaddling
"Newborn Stress Scale" | After the massage
"Newborn Stress Scale" | After the swaddling

SECONDARY OUTCOMES:
Baby's heart rate | A minutes before massage
Baby's respiratory rate | A minutes before massage
Baby's oxygen saturation | A minutes before massage
Baby's body temperature | A minutes before massage
Baby's heart rate | 5th minute of the massage
Baby's respiratory rate | 5th minute of the massage
Baby's oxygen saturation | 5th minute of the massage
Baby's body temperature | 5th minute of the massage
Baby's heart rate | A minutes after massage
Baby's respiratory rate | A minutes after massage
Baby's oxygen saturation | A minutes after massage
Baby's body temperature | A minutes after massage
Baby's heart rate | A minutes before swaddling
Baby's respiratory rate | A minutes before swaddling
Baby's oxygen saturation | A minutes before swaddling
Baby's body temperature | A minutes before swaddling
Baby's heart rate | In the fifth minute of the swaddling
Baby's respiratory rate | 5th minute of the swaddling
Baby's oxygen saturation | 5th minute of the swaddling
Baby's body temperature | 5th minute of the swaddling
Baby's heart rate | A minutes after swaddling
Baby's respiratory rate | A minutes after swaddling
Baby's oxygen saturation | A minutes after swaddling
Baby's body temperature | A minutes after swaddling

CONTACTS AND LOCATIONS:
Overall Officials: Hatice BAL YILMAZ, Prof., Study Director — Ege University; Pınar DOGAN, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No